CLINICAL TRIAL: NCT04005326
Title: Quadratus Lumborum Block Versus Fascia Iliaca Block for Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block Versus Fascia Iliaca Block for Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassant M. Abdelhamid (Other)
Responsible Party: Sponsor-Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-144-2018
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB Group (Experimental): this group will receive ultrasound-guided transmuscular quadratus lumborum block; (Anterior QLB or QLB III)
  Interventions: Procedure: quadratus lumborum block; (Anterior QLB or QLB III); Procedure: Subarachnoid block
- FIB Group (Experimental): this group will receive suprainguinal fascia iliaca block
  Interventions: Procedure: suprainguinal fascia iliaca block; Procedure: Subarachnoid block

INTERVENTIONS:
Procedure: quadratus lumborum block; (Anterior QLB or QLB III) — The patient will be in the lateral position. A low frequency convex probe will be vertically attached above the iliac crest and a needle will be inserted in plane from the posterior edge of the convex probe through the quadratus lumborum in an anteromedial direction. The needle tip will be placed between the psoas major muscle and the quadratus lumborum muscle. After negative aspiration, 30 mL of 0.25 % of bupivacaine will be injected into the fascial plane incrementally, aspirating every 5 ml.
  Arms: QLB Group
Procedure: suprainguinal fascia iliaca block — In supine position, a high frequency linear probe will be placed in the inguinal crease. Scan starting laterally from the femoral artery and nerve in inguinal crease to identify the sartorius muscle, tracing the muscle until it's origin to anterior superior iliac spine. The shadow of the bony of iliac crest & iliacus muscle will be seen, the end point of the injection is deep to the fascia iliaca and above the iliacus muscle in the lateral part of the iliacus muscle. After negative aspiration, 30 mL of 0.25 % of bupivacaine will be injected under the fascial plane incrementally, aspirating every 5 ml.
  Arms: FIB Group
Procedure: Subarachnoid block — Patients will receive SAB using 25g spinal needle in the lateral position. Fifteen milligrams of hyperbaric bupivacaine will be administered at L3-L4 or at L4-L5 interspace in addition to 25 mcg fentanyl with rapid crystalloid co-load.
  Spinal anesthesia will be considered successful when a bilateral block to T12, as assessed by loss of cold (cold ice) and pain (a 23-gauge needle) sensations, will be established 10 -minutes after the intrathecal injection. If spinal anesthesia failed, such patients will be administered general anesthesia and will be excluded from this study.
  Other Names: spinal anesthesia

SUMMARY:
Quadratus lumborum block is a newly developed block with good performance in lower abdominal surgery. In a cadaveric study, the spread of local anesthetic in the anterior approach of QL block (QL3) was reported to cover nerve roots from T10 to L3. Thus, it was hypothesized that this approach could be used in hip surgeries with minimal motor affection.

This study aims to compare QL3 block and suprainguinal Fascia Iliaca block in the duration of postoperative analgesia, pain scores, motor power in quadriceps muscle, and side effects.

DETAILED DESCRIPTION:
A randomized, controlled, double blinded, trial will be conducted in Cairo university hospital. Written informed consent will be obtained from all participants. Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes. Patients scheduled for hip replacement surgeries under subarachnoid block (SAB). e.g. hip hemiarthroplasty, total hip arthroplasty.

On arrival of the patients to regional anesthesia room, patients will be secured with 18-gauge intravenous cannula, and will receive ondansetron (4 mg), and dexamethasone (8 mg IV). Monitoring will include Electrocardiography, non-invasive arterial blood pressure, and pulse oximetry.

Before receiving subarachinoid block, patients will be randomly assigned into one of the two study groups:

QLB Group (n=17): this group will receive ultrasound-guided transmuscular quadratus lumborum block; (Anterior QLB or QLB III) FIB Group (n=17): this group will receive suprainguinal fascia iliaca block To achieve double blinding, patients will receive the block with 30 mL bupivacaine (0.25%) by the anesthetist. Another doctor not involved in the block procedure will evaluate the patients postoperative.

After finishing the block & assessment of motor power of quadriceps femoris muscle , patient will receive midazolam (2mg intravenous), and then transferred to operation room.

Postoperatively, all patients will receive 1 g paracetamol every 6 hours and 30 mg ketorolac every 12 hours.

If the visual analogue scale (VAS) is 4 or more, a 2 mg morphine increment will be added per time to maintain a resting VAS at <3 with maximum total 24-hours morphine 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip replacement surgeries under subarachnoid block (SAB). e.g. hip hemiarthroplasty, total hip arthroplasty.

Exclusion Criteria:

* Coagulopathy, infection at the injection site,.
* Allergy to local anesthetics.
* Severe cardiopulmonary disease (≥ASA IV),.
* Diabetic or other neuropathies.
* Patients receiving opioids for chronic analgesic therapy.
* Contraindication to spinal anesthesia.
* Inability to comprehend visual analogue scale (VAS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-10-05 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours postoperative
  If the visual analogue scale (VAS) is 4 or more, a 2 mg morphine increment will be added per time to maintain a resting VAS at <3 with maximum total 24-hours morphine 10 mg.

SECONDARY OUTCOMES:
Static visual analogue pain scale | 24 hours postoperative
  Visual analogue pain scale (VAS) at rest. The pain visual analogue pain scale( VAS) is a continuous scale 10 centimeters (100 mm) in length. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).
Dynamic visual analogue pain scale | 24 hours postoperative
  Visual analogue pain scale (VAS) on movement. The pain visual analogue pain scale( VAS) is a continuous scale 10 centimeters (100 mm) in length. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).
Onset of sensory block of quadratus lumborum block and fascia iliaca block | 30 minutes
  the time interval between the injection of the study medication till complete loss of sensation
Time to first postoperative analgesic request | 24 hours postoperative
  morphine increment will be added per time to maintain a resting VAS at <3 with maximum
Total morphine requirements | 24 hours postoperative
  If the visual analogue scale (VAS) is 4 or more, a 2 mg morphine increment will be added per time to maintain a resting VAS at <3 with maximum total 24-hours morphine 10 mg.
Assessment of the quadriceps muscle power. | 24 hours
  the patient will be in supine position and the patient's knee will be fully flexed, and the patient will be asked to extend it. The motor block is classified as follows: grade 0; normal muscle power, grade I; motor weakness, grade II; complete motor paralysis
Time needed to perform the block | 30 minutes
  the total time of the procedure (quadratus lumborum block or fascia iliaca block) started from patient positioning till completion of local anesthesia injection.
incidence of pain during positioning for spinal block | 30 minutes
  to assess the ability of either two types of the the blocks to relieve pain during positioning for spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Hasanin, M.D., Principal Investigator — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullock WM, Yalamuri SM, Gregory SH, Auyong DB, Grant SA. Ultrasound-Guided Suprainguinal Fascia Iliaca Technique Provides Benefit as an Analgesic Adjunct for Patients Undergoing Total Hip Arthroplasty. J Ultrasound Med. 2017 Feb;36(2):433-438. doi: 10.7863/ultra.16.03012. Epub 2016 Dec 10. PMID 27943417
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Bang S, Chung J, Jeong J, Bak H, Kim D. Efficacy of ultrasound-guided fascia iliaca compartment block after hip hemiarthroplasty: A prospective, randomized trial. Medicine (Baltimore). 2016 Sep;95(39):e5018. doi: 10.1097/MD.0000000000005018. PMID 27684871
- [Derived] Nassar H, Hasanin A, Sewilam M, Ahmed H, Abo-Elsoud M, Taalab O, Rady A, Zoheir HA. Transmuscular Quadratus Lumborum Block versus Suprainguinal Fascia Iliaca Block for Hip Arthroplasty: A Randomized, Controlled Pilot Study. Local Reg Anesth. 2021 Apr 20;14:67-74. doi: 10.2147/LRA.S308964. eCollection 2021. PMID 33907462